CLINICAL TRIAL: NCT05874661
Title: The Effect of Focus of Attention on Motor Performance and Learning During a Sit to Stand Task in Individuals Post-stroke
Brief Title: FOA on Sit to Stand in Individuals Post Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western Carolina University (Other)
Collaborators: Mission Health System, Asheville, NC (Other); Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: WesternCarolinaU; Full PhD Dissertation Study (Other: WCU)
Record Dates: First submitted 2023-03-29; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Stroke, Acute
Keywords: Focus of Attention; Motor Learning; Sit to Stand
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: This study will be a randomized cross over study. Individuals will be randomized into either an internal or external focus condition for the first week of the study and be crossed over to the other condition in the second week.
Who Masked: Participant
Masking Description: Participants will not be aware of their group allocation compared to the other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internal Focus of Attention Group (Active Comparator): Participants will be given instructions that make them think about their body's movements.
  Participants assigned to this condition first will complete the external focus condition second in the cross over.
  Interventions: Other: Internal Focus of Attention
- Extneral Focus of Attention Group (Experimental): Participants will be given instructions that make them think about an outside target or outcome.
  Participants assigned to this condition first will complete the internal focus condition second in the cross over.
  Interventions: Other: External Focus of Attention

INTERVENTIONS:
Other: External Focus of Attention — Focus of attention refers to what a person is thinking about during a task, with an external focus being thinking about a target or outcome in the environment.
  Arms: Extneral Focus of Attention Group
Other: Internal Focus of Attention — Focus of attention refers to what a person is thinking about during a task, with an internal focus being thinking about what one's body is doing.
  Arms: Internal Focus of Attention Group

SUMMARY:
Focus of attention refers to what a person is thinking about during a task, with an internal focus being thinking about what one's body is doing and an external focus being thinking about a target or outcome in the environment. The purpose of this study is to fill some of the gaps in the literature by examining the effects of focus of attention on performance and learning of sit to stand in individuals post stroke. This study will investigate whether an internal or external focus of attention can lead to improved use of the affected lower extremity during the sit to stand transition, while maintaining an upright trunk position.

DETAILED DESCRIPTION:
Introduction More than 795,000 people have a stroke in the United States each year, one every 40 seconds, leading to 7.6 million Americans who have had a stroke. Further, stroke remains the leading cause of long term disability, with greater than 50 percent of stroke survivors being chronically disabled. One factor contributing to disability is the difficulty with sit to stand transfers.

Individuals post stroke present with decreased knee moment on the affected side resulting in a less efficient sit to stand transition. In addition, individuals post stroke demonstrate increased trunk displacement in the mediolateral direction towards the unaffected side and weight distribution asymmetry. Cheng et al. found that individuals post stroke who were classified as fallers took more time to stand, had more mediolateral sway, and pushed less force through the affected lower extremity during sit to stand.

Sit to stand training is essential during rehabilitation post stroke to improve the ability to stand with a more normal biomechanical pattern and to positively impact other aspects of mobility. Several studies underline the importance of sit to stand training with a focus on increasing use of the affected lower extremity. Forced use training of the affected lower extremity has led to increased muscle activity in the affected limb, improved balance, gait kinematics, gait symmetry, gait velocity, and quality of life.

In order to make sit to stand training more effective the type of instruction and feedback is key. Based on a number of studies, simply changing two to three words of instruction can lead to more effective outcomes. This impactful change in instruction is based on focus of attention research, exploring the difference between internal and external focus instruction. An internal focus refers to thinking about one's own body movements, while an external focus is focusing on an outcome or impact on the environment. An example of internal focus is thinking about what one's shoulders or arm is doing while shooting a basketball, while an external focus would be thinking about the effect on the ball or the basket. Over 80 studies have supported an external focus being more effective than an internal focus of attention in the healthy adult and sports population.

The research in the stroke population related to focus of attention is sparse and contradictory. Some studies show an external focus being detrimental to movement fluency, while others find that an external focus leads to better outcomes. The remaining studies in the stroke population, however, have found no difference between internal and external foci. Most of these studies examined the effect of attentional focus during practice but did not include retention testing, thus the effects on motor learning have not been assessed. In addition, these studies have not examined the effects of focus of attention on functional movements such as sit to stand.

Individuals post stroke may respond differently to focus of attention compared to healthy adults due to their impairments and cerebral changes. Individuals post stroke can have decreased executive function including information processing. Also, these individuals may lose some motor automaticity leading them to consciously try to control their movement.

Statement of the Problem Impairments following stroke often lead to functional limitations such as difficulty performing a sit to stand transfer, which may affect independence in other activities of daily living. Individuals following stroke often perform sit to stand transfers less efficiently than individuals without stroke. This inefficiency is due in part to asymmetry between the unaffected and affected lower extremity. Training people to use the affected side more may increase efficiency of their movement and decrease fall risk. The type of instruction and feedback, specifically focus of attention instruction, may impact how well people following stroke learn to use the affected side more during sit to stand transfers. At this time, the effect of focus of attention instruction and feedback on the increased use of the affected side during sit to stand in individuals post stroke is unknown.

Purpose The purpose of this study is to fill some of the gaps in the literature by examining the effects of focus of attention on performance and learning of sit to stand in individuals post stroke. This study will investigate whether an internal or external focus of attention can lead to improved use of the affected lower extremity during the sit to stand transition, while maintaining an upright trunk position.

Research Questions

The following research questions will be addressed in this study:

1. Does an internal or external focus enhance motor learning of a sit to stand task in which learning will be evaluated using a retention and transfer test? Retention will refer to the ability to perform the sit to stand task without explicit instruction five minutes and one hour after practice. Transfer of learning will be evaluated by exploring the effects of sit to stand training on gait symmetry.
2. Does an internal or external focus lead to an improved performance of a sit to stand task during training as measured by an increased weight shift towards the affected side and upright trunk alignment?

Participant demographics and clinical information will be collected, including age, gender, weight, height, location of stroke, how long ago the stroke occurred, and fall history. All participants will consent to participation in this study. The Star Cancellation Test and Montreal Cognitive Assessment (MOCA) will be used to determine eligibility. Gait speed and the Fugl Meyer for the lower extremity, excluding reflexes, will also be completed to help describe the sample. Blood pressure, heart rate, and oxygen saturation, via a pulse oximeter, will be taken and a gait belt will be placed on the participant prior to the start of baseline measures. Temporospatial gait parameters will be collected using the GAITRite mat at baseline, 5 minutes after training, and 1 hour after training. Temporospatial gait parameters will be averaged across four passes over the GAITRite mat at each measurement session. Participants will be instructed to 'walk past the end of the mat at your normal comfortable pace'. Gait speed will be recorded at baseline as part of the individuals' baseline measurements.

Participants will then be seated on a hi-lo table with their feet on the HR pressure mat for baseline assessment of sit to stand. Initial mat height will be determined by raising or lowering the mat table until the femur is parallel to the floor. This initial mat position will be the height used during each reassessment at baseline, 5 minutes after training, and 1 hour post training. This height will also be used to decide the mat positions needed during training. After the initial mat height is achieved and recorded, an IMU marker will be placed on the superior third of the sternum directly inferior to the sternal notch.

Next, participants will be asked to stand up and sit down to determine comfortable foot placement in relation to their knees. Tape marks will be placed in front of the toes and on the lateral edges of both feet as well as around the buttocks to allow for a standardized starting position for all assessment timepoints. For all data collection during baseline, 5 minutes post, and 1 hour post training, participants will be instructed to "please stand up three times at your normal speed without your arms if possible". The average force under the affected foot and the average overall force beneath both feet during the sit to stand transition will be captured by the HR pressure mat. The maximal lateral trunk position will be captured throughout this transition by the IMU marker. If individuals need to use their upper extremities this will be recorded.

After baseline data collection, participants will be randomized into either the internal or external focus condition. Initial group allocation will be determined by a random number generator, blocks of 6 with a 1:1 ratio. Group allocation envelops will be opened directly prior to acquisition trials so baseline assessors will be blinded to group assignment of participants. Participants will be blinded to initial group assignment throughout the entirety of the sessions.

Training Prior to training, a demonstration of the task will be provided to the participants. Those in the external focus condition will be told, "as you stand up and as you sit down try to bring the targets together like this". Those in the internal focus condition will be told, "as you stand up and as you sit down bring your right/left (R/L) shoulder and R/L hip as far to the R/L as possible." Participants will be asked to perform one repetition with the question "can you show me?". The demonstration is only provided before the first set but these same instructions will be given prior to the start of each successive set during training.

During training trials, individuals will perform four sets of ten sit to stand repetitions. During the external focus condition, foam circles will be taped to the participant's lateral shoulder and lateral hip. In order to define this distance, participant girth will be measured in a seated position, by measuring the distance between bilateral outer thighs, using greater trochanters as landmarks. When the individual is standing in midline targets will be placed half of this girth measurement plus 10 centimeters away from the lateral tip of their acromion and another target placed the same distance away from their greater trochanter.

During training, participants will perform four sets of sit to stand transitions with the mat at progressively lower seat heights to increasingly challenge the participants, with instruction and feedback consistent with their condition allocation. The four sets will occur in the following sequences: 130 percent of the initial mat height determined at baseline assessment, 120 percent, 110 percent and 100 percent. Each set will end after the tenth repetition or when the participant reports a RPE rating of >15/20. If participants are unable to complete 10 repetitions, the number completed will be recorded for each trial. Two minute rest breaks will occur between each set or until the participant reports a rate of perceived exertion (RPE) of <12/20 on the Borg RPE scale. During training, one verbal correction will be given during each set after the 2nd, 4th, and 7th trials, based on patient performance and condition allocation. The feedback provided will be recorded.

Immediately after the training, participants will take a 5 minute break followed by the post-5 minute retention test in which instrumented sit to stand and gait will be administered. Following the retention test, individuals will complete a general health questionnaire. Approximately one hour after the training ends, 1-hour retention testing will be administered consisting of 3 instrumented sit to stands and gait over the GAITRite. After the immediate long term data collection, the participants will complete the post manipulation questionnaire to determine what the participants were focusing on during training.

One week later participants will return and complete the same protocol in the opposite attentional condition to which they were initially randomized.

ELIGIBILITY:
Inclusion Criteria:

* post stroke <6 months
* at least 18 years of age, of any gender, race, or ethnic group

Exclusion Criteria:

* Unable to stand unassisted from a standard height, 20" chair, with or without upper extremity assistance
* Unable to ambulate 20 feet without physical assistance or
* Moderate to severely impaired cognition with a score of <10/30 on the Montreal Cognitive Assessment (MOCA)
* Contraversive pushing with >1 according to the Scale for Contraversive Pushing Scale
* Neglect as evidenced by <44/56 on the Star Cancellation Test
* Any orthopedic or other neurologic conditions that impact their ability to transition from sit to stand

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-04-02 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of force under affected lower extremity | Baseline
  HR Pressure mat - Symmetry under the feet will be measured using a 61.26 X 58.72 cm pedobarograph with a 48.8 X 44.7 cm active sensing area during the sit to stand transition. The mat has 3.9 sensors/cm2 with a 185 Hz scanning rate. The mat will be calibrated prior to the start of the study.
Proportion of force under affected lower extremity | Acquisition (one 1 hour training)
  HR Pressure mat - Symmetry under the feet will be measured using a 61.26 X 58.72 cm pedobarograph with a 48.8 X 44.7 cm active sensing area during the sit to stand transition. The mat has 3.9 sensors/cm2 with a 185 Hz scanning rate. The mat will be calibrated prior to the start of the study.
Proportion of force under affected lower extremity | Short term (5 minutes after training)
  HR Pressure mat - Symmetry under the feet will be measured using a 61.26 X 58.72 cm pedobarograph with a 48.8 X 44.7 cm active sensing area during the sit to stand transition. The mat has 3.9 sensors/cm2 with a 185 Hz scanning rate. The mat will be calibrated prior to the start of the study.
Proportion of force under affected lower extremity | Long term (1 hour after training)
  HR Pressure mat - Symmetry under the feet will be measured using a 61.26 X 58.72 cm pedobarograph with a 48.8 X 44.7 cm active sensing area during the sit to stand transition. The mat has 3.9 sensors/cm2 with a 185 Hz scanning rate. The mat will be calibrated prior to the start of the study.
Trunk alignment | Baseline
  IMU sensors -One Delsys inertial measurement units (IMUs) will be placed on the sternum just inferior to the sternal notch to capture vertical trunk alignment throughout sit to stand.
Trunk alignment | Acquisition (1 hour training)
  IMU sensors -One Delsys inertial measurement units (IMUs) will be placed on the sternum just inferior to the sternal notch to capture vertical trunk alignment throughout sit to stand.
Trunk alignment | Short term (5 minutes post training)
  IMU sensors -One Delsys inertial measurement units (IMUs) will be placed on the sternum just inferior to the sternal notch to capture vertical trunk alignment throughout sit to stand.
Trunk alignment | Long term (1 hour post training)
  IMU sensors -One Delsys inertial measurement units (IMUs) will be placed on the sternum just inferior to the sternal notch to capture vertical trunk alignment throughout sit to stand.
Gait symmetry | Baseline
  GaitRite - A 20'X 4' GAITRite will be used to gather gait speed and analyze spatial temporal aspects of gait. The GAITRite mat is an electronic walkway which uses pressure activated sensors to map out foot placement during gait using a quadrilateral blocking system. The walkway is made up of sensor pads, each of which has 2,304 sensors arranged in 48X48 grids. The measurements are provided using x,y coordinates and algorithms in the computer system use this information to group sensors into footprints. The mat has a spatial resolution of 1.27 cm and a spatial resolution accuracy of 1.27 cm. The mat will be set at 120 Hz sampling rate. All other parameters are fixed. GAITRite software will be used to collect percent of time spent in affected lower extremity stance compared to total stance time.
Gait symmetry | Short term (5 minutes after training)
  GaitRite - A 20'X 4' GAITRite will be used to gather gait speed and analyze spatial temporal aspects of gait. The GAITRite mat is an electronic walkway which uses pressure activated sensors to map out foot placement during gait using a quadrilateral blocking system. The walkway is made up of sensor pads, each of which has 2,304 sensors arranged in 48X48 grids. The measurements are provided using x,y coordinates and algorithms in the computer system use this information to group sensors into footprints. The mat has a spatial resolution of 1.27 cm and a spatial resolution accuracy of 1.27 cm. The mat will be set at 120 Hz sampling rate. All other parameters are fixed. GAITRite software will be used to collect percent of time spent in affected lower extremity stance compared to total stance time.
Gait symmetry | Long term (1 hour after training)
  GaitRite - A 20'X 4' GAITRite will be used to gather gait speed and analyze spatial temporal aspects of gait. The GAITRite mat is an electronic walkway which uses pressure activated sensors to map out foot placement during gait using a quadrilateral blocking system. The walkway is made up of sensor pads, each of which has 2,304 sensors arranged in 48X48 grids. The measurements are provided using x,y coordinates and algorithms in the computer system use this information to group sensors into footprints. The mat has a spatial resolution of 1.27 cm and a spatial resolution accuracy of 1.27 cm. The mat will be set at 120 Hz sampling rate. All other parameters are fixed. GAITRite software will be used to collect percent of time spent in affected lower extremity stance compared to total stance time.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley W Hyatt, DPT, PhD (C), Principal Investigator — Western Carolina University
Locations (2):
- United States (2):
  - CarePartners, Asheville, North Carolina
  - Western Carolina University, Cullowhee, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided
Open to sharing data upon request and approval of IRB at Mission Health

REFERENCES:
- [Background] Abdullahi A, Truijen S, Umar NA, Useh U, Egwuonwu VA, Van Criekinge T, Saeys W. Effects of Lower Limb Constraint Induced Movement Therapy in People With Stroke: A Systematic Review and Meta-Analysis. Front Neurol. 2021 Mar 23;12:638904. doi: 10.3389/fneur.2021.638904. eCollection 2021. PMID 33833730
- [Background] CIR Sytems. (2013). GAITRite Electronic Walkway Technical Reference. Technical Reference (WI-02-15), 1-50.
- [Background] Matscan, F. (2021). Footmat TM user manual 7.1x.
- [Background] Orrell AJ, Masters RS, Eves FF. Reinvestment and movement disruption following stroke. Neurorehabil Neural Repair. 2009 Feb;23(2):177-83. doi: 10.1177/1545968308317752. Epub 2008 Nov 5. PMID 18987385
- [Result] Aloraini SM, Glazebrook CM, Pooyania S, Sibley KM, Singer J, Passmore S. An external focus of attention compared to an internal focus of attention improves anticipatory postural adjustments among people post-stroke. Gait Posture. 2020 Oct;82:100-105. doi: 10.1016/j.gaitpost.2020.08.133. Epub 2020 Aug 29. PMID 32911092
- [Result] Billinger SA, Guo LX, Pohl PS, Kluding PM. Single limb exercise: pilot study of physiological and functional responses to forced use of the hemiparetic lower extremity. Top Stroke Rehabil. 2010 Mar-Apr;17(2):128-39. doi: 10.1310/tsr1702-128. PMID 20542855
- [Result] Cheng PT, Liaw MY, Wong MK, Tang FT, Lee MY, Lin PS. The sit-to-stand movement in stroke patients and its correlation with falling. Arch Phys Med Rehabil. 1998 Sep;79(9):1043-6. doi: 10.1016/s0003-9993(98)90168-x. PMID 9749681
- [Result] Durham KF, Sackley CM, Wright CC, Wing AM, Edwards MG, van Vliet P. Attentional focus of feedback for improving performance of reach-to-grasp after stroke: a randomised crossover study. Physiotherapy. 2014 Jun;100(2):108-15. doi: 10.1016/j.physio.2013.03.004. Epub 2013 Jun 21. PMID 23796803
- [Result] Fasoli SE, Trombly CA, Tickle-Degnen L, Verfaellie MH. Effect of instructions on functional reach in persons with and without cerebrovascular accident. Am J Occup Ther. 2002 Jul-Aug;56(4):380-90. doi: 10.5014/ajot.56.4.380. PMID 12125827
- [Result] Hsu CJ, Kim J, Roth EJ, Rymer WZ, Wu M. Forced Use of the Paretic Leg Induced by a Constraint Force Applied to the Nonparetic Leg in Individuals Poststroke During Walking. Neurorehabil Neural Repair. 2017 Dec;31(12):1042-1052. doi: 10.1177/1545968317740972. Epub 2017 Nov 16. PMID 29145773
- [Result] Kal EC, van der Kamp J, Houdijk H, Groet E, van Bennekom CA, Scherder EJ. Stay Focused! The Effects of Internal and External Focus of Attention on Movement Automaticity in Patients with Stroke. PLoS One. 2015 Aug 28;10(8):e0136917. doi: 10.1371/journal.pone.0136917. eCollection 2015. PMID 26317437
- [Result] Kal E, Houdijk H, van der Kamp J, Verhoef M, Prosee R, Groet E, Winters M, van Bennekom C, Scherder E. Are the effects of internal focus instructions different from external focus instructions given during balance training in stroke patients? A double-blind randomized controlled trial. Clin Rehabil. 2019 Feb;33(2):207-221. doi: 10.1177/0269215518795243. Epub 2018 Aug 31. PMID 30168348
- [Result] Katzan, I. L. (2013). Epidemiology of stroke. Handbook of Clinical Nutrition and Stroke, 3-14. https://doi.org/10.1007/978-1-62703-380-0_1
- [Result] Kim GJ, Hinojosa J, Rao AK, Batavia M, O'Dell MW. Randomized Trial on the Effects of Attentional Focus on Motor Training of the Upper Extremity Using Robotics With Individuals After Chronic Stroke. Arch Phys Med Rehabil. 2017 Oct;98(10):1924-1931. doi: 10.1016/j.apmr.2017.06.005. Epub 2017 Jun 24. PMID 28652064
- [Result] Lopez AD, Mathers CD, Ezzati M, Jamison DT, Murray CJ. Global and regional burden of disease and risk factors, 2001: systematic analysis of population health data. Lancet. 2006 May 27;367(9524):1747-57. doi: 10.1016/S0140-6736(06)68770-9. PMID 16731270
- [Result] Muckel S, Mehrholz J. Immediate effects of two attention strategies on trunk control on patients after stroke. A randomized controlled pilot trial. Clin Rehabil. 2014 Jul;28(7):632-6. doi: 10.1177/0269215513513963. Epub 2014 Jan 22. PMID 24452700
- [Result] Patterson KK, Parafianowicz I, Danells CJ, Closson V, Verrier MC, Staines WR, Black SE, McIlroy WE. Gait asymmetry in community-ambulating stroke survivors. Arch Phys Med Rehabil. 2008 Feb;89(2):304-10. doi: 10.1016/j.apmr.2007.08.142. PMID 18226655
- [Result] Tsao CW, Aday AW, Almarzooq ZI, Alonso A, Beaton AZ, Bittencourt MS, Boehme AK, Buxton AE, Carson AP, Commodore-Mensah Y, Elkind MSV, Evenson KR, Eze-Nliam C, Ferguson JF, Generoso G, Ho JE, Kalani R, Khan SS, Kissela BM, Knutson KL, Levine DA, Lewis TT, Liu J, Loop MS, Ma J, Mussolino ME, Navaneethan SD, Perak AM, Poudel R, Rezk-Hanna M, Roth GA, Schroeder EB, Shah SH, Thacker EL, VanWagner LB, Virani SS, Voecks JH, Wang NY, Yaffe K, Martin SS. Heart Disease and Stroke Statistics-2022 Update: A Report From the American Heart Association. Circulation. 2022 Feb 22;145(8):e153-e639. doi: 10.1161/CIR.0000000000001052. Epub 2022 Jan 26. PMID 35078371
- [Result] Onursal Kilinc O, De Ridder R, Kilinc M, Van Bladel A. Trunk and lower extremity biomechanics during sit-to-stand after stroke: A systematic review. Ann Phys Rehabil Med. 2023 Apr;66(3):101676. doi: 10.1016/j.rehab.2022.101676. Epub 2022 Dec 5. PMID 35597449
- [Result] Virani SS, Alonso A, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Shay CM, Spartano NL, Stokes A, Tirschwell DL, VanWagner LB, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2020 Update: A Report From the American Heart Association. Circulation. 2020 Mar 3;141(9):e139-e596. doi: 10.1161/CIR.0000000000000757. Epub 2020 Jan 29. PMID 31992061
- [Result] Wu M, Hsu CJ, Kim J. Forced use of paretic leg induced by constraining the non-paretic leg leads to motor learning in individuals post-stroke. Exp Brain Res. 2019 Oct;237(10):2691-2703. doi: 10.1007/s00221-019-05624-w. Epub 2019 Aug 12. PMID 31407027
- [Result] Wulf, G. (2013). Attentional focus and motor learning: A review of 15 years. International Review of Sport and Exercise Psychology, 6(1), 77-104. https://doi.org/10.1080/1750984X.2012.723728
- [Result] Wulf G, McNevin N, Shea CH. The automaticity of complex motor skill learning as a function of attentional focus. Q J Exp Psychol A. 2001 Nov;54(4):1143-54. doi: 10.1080/713756012. PMID 11765737
- [Result] Yu WH, Liu WY, Wong AM, Wang TC, Li YC, Lien HY. Effect of forced use of the lower extremity on gait performance and mobility of post-acute stroke patients. J Phys Ther Sci. 2015 Feb;27(2):421-5. doi: 10.1589/jpts.27.421. Epub 2015 Feb 17. PMID 25729182
- [Result] Zinn S, Bosworth HB, Hoenig HM, Swartzwelder HS. Executive function deficits in acute stroke. Arch Phys Med Rehabil. 2007 Feb;88(2):173-80. doi: 10.1016/j.apmr.2006.11.015. PMID 17270514